CLINICAL TRIAL: NCT02667873
Title: A Phase 1 Trial of SL-801, a Novel Inhibitor of XPO1 Nuclear Export, in Patients With Advanced Solid Tumors
Brief Title: A Trial of a Novel XPO1 Inhibitor in Participants With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stemline Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STML-801-0115
Record Dates: First submitted 2015-11-03; First posted 2016-01-29 (Estimated); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SL-801 (Experimental): The starting dose regimen of SL-801 (that is, the dose regimen in Cohort 1) is 5 milligrams (mg)/day on Days 1-4 and 8-11 every 21 days. In the second portion of the dose escalation stage, participants receive SL-801 orally once daily on days 1-2, 8-9, 15-16 and 22-23 every 28 days. The starting dose will be 70 mg/day (the next planned dose level). The SL-801 dose regimen for a particular participant is dependent on the cohort in which the participant is enrolled.
  Interventions: Drug: SL-801

INTERVENTIONS:
Drug: SL-801 — SL-801 is a small-molecule inhibitor of the nuclear export protein Exportin-1 (XPO1).
  Other Names: Felezonexor

SUMMARY:
Study SL-801-0115 is a dose-escalation study evaluating multiple doses and schedules of orally administered SL-801 in participants with advanced solid tumors.

DETAILED DESCRIPTION:
Study SL-801-0115 is a first-in-human, dose-escalation study in participants with advanced (that is, metastatic or locally advanced and unresectable) solid tumors that are resistant to or relapsed following available standard systemic therapy or for which there is no standard systemic therapy and additional radiation therapy, or other loco-regional therapies are not considered feasible. Eligible participants will be enrolled and receive treatment with SL-801. SL-801 will be administered orally, and the dose regimen will depend on the cohort in which the participant is enrolled.

The study plans to enroll approximately 70 adult participants at multiple study centers in the United States.

ELIGIBILITY:
Inclusion Criteria:

* The participant must have histologic or cytologic evidence of a malignant solid tumor and must have disease that is resistant to or relapsed following available standard systemic therapy, or for which there is no standard systemic therapy or reasonable therapy likely to result in clinical benefit.
* The participant must have advanced disease, defined as cancer that is either metastatic, or locally advanced and unresectable (and for which additional radiation therapy or other locoregional therapies are not considered feasible).
* The participant must have disease that is measurable by standard imaging techniques, per the Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST 1.1), or evaluable per RECIST 1.1. (For participants with prior radiation therapy, measurable lesions must be outside of any prior radiation field[s], unless disease progression has been documented at that disease site subsequent to radiation.)
* The participant is ≥18 years old.
* The participant has an Eastern Cooperative Oncology Group Performance Status of 0-2.
* The participant has adequate baseline organ function, as demonstrated by the following:

  * Serum creatinine ≤1.5 × institutional upper limit of normal (ULN) or calculated creatinine clearance >30 milliliters (mL)/minute.
  * Serum albumin ≥2.5 grams/deciliter (g/dL).
  * Bilirubin ≤1.5 × institutional ULN.
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 × institutional ULN (participants with hepatic metastases must have AST/ALT ≤5 times ULN).
  * International normalized ratio ≤1.5 or prothrombin time ≤1.5 × ULN; and either partial thromboplastin time or activated partial thromboplastin time (partial thromboplastin time or activated partial thromboplastin time) ≤1.5 × ULN.
* The participant has adequate baseline hematologic function, as demonstrated by the following:

  * Absolute neutrophil count ≥1.5×10^9/liter (L)
  * Hemoglobin ≥8 g/dL, with no red blood cell transfusions within the prior 14 days.
  * Platelet count ≥100×10^9/L, with no platelet transfusions within the prior 14 days.
* If the participant is a woman of childbearing potential, she has had a negative serum or urine pregnancy test within 1 week prior to treatment.
* The participant (male and female) agrees to use acceptable contraceptive methods for the duration of time on the study and continue to use acceptable contraceptive methods for 1 month after the last dose of SL-801.
* The participant has signed informed consent prior to initiation of any study-specific procedures or treatment.
* The participant is able to adhere to the study visit schedule and other protocol requirements, including follow-up for survival assessment.

Exclusion Criteria:

* The participant has persistent clinically significant ≥Grade 2 toxicities from previous anticancer therapy (excluding Grade 2 chemotherapy-related neuropathy which is permitted, and excluding Grade 2-3 laboratory abnormalities if they are not associated with symptoms, are not considered clinically significant by the Investigator, and can be managed with available medical therapies).
* The participant has received treatment with chemotherapy, external-beam radiation, or other systemic anticancer therapy within 28 days prior to study entry (Participants with advanced prostate cancer who are receiving luteinizing hormone releasing hormone [LHRH] agonists are permitted onto the study and should continue use of these agents during study treatment).
* The participant has received treatment with an investigational systemic anticancer agent within 28 days prior to C1D1.
* The participant has previously received treatment with SL-801 or another investigational agent that inhibits the XPO1/CRM1 pathway.
* The participant has an additional active malignancy that may confound the assessment of the study endpoints. Participants with a past cancer history (active malignancy within 2 years prior to study entry) with substantial potential for recurrence must be discussed with the Sponsor before study entry. Participants with the following concomitant neoplastic diagnoses are eligible: non-melanoma skin cancer, carcinoma in situ (including transitional cell carcinoma, cervical intraepithelial neoplasia), organ-confined prostate cancer with no evidence of progressive disease.
* The participant has clinically significant cardiovascular disease (for example, uncontrolled or any New York Heart Association Class 3 or 4 congestive heart failure, uncontrolled angina, history of myocardial infarction, unstable angina or stroke within 6 months prior to study entry, uncontrolled hypertension or clinically significant arrhythmias not controlled by medication).
* The participant has uncontrolled, clinically significant pulmonary disease (for example, chronic obstructive pulmonary disease, pulmonary hypertension) that, in the Investigator's opinion, would put the participant at significant risk for pulmonary complications during the study.
* The participant has known active or suspected brain or leptomeningeal metastases. (Central nervous system [CNS] imaging is not required prior to study entry unless there is a clinical suspicion of CNS involvement). Participants with stable, treated brain metastases are eligible provided there is no evidence of CNS disease growth on imaging for at least 3 months following radiation therapy or other locoregional ablative therapy to the CNS.
* The participant is receiving immunosuppressive therapy for prophylaxis following a prior organ transplant (solid organ or allogeneic stem cell) or management of immune-mediated toxicities due to immunotherapy. Low-dose corticosteroid (defined as < 10 mg/day of prednisone or equivalent) therapy is permitted.
* The participant has uncontrolled intercurrent illness including, but not limited to, uncontrolled infection, disseminated intravascular coagulation, or psychiatric illness/social situations that would limit compliance with study requirements.
* The participant is pregnant or breast feeding.
* The participant has known positive status for human immunodeficiency virus active or chronic Hepatitis B or Hepatitis C.
* The participant is oxygen dependent.
* The participant has any medical condition which in the opinion of the Investigator places the patient at an unacceptably high risk for toxicities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2016-02-23 (Actual); Primary Completion 2021-10-06 (Actual); Study Completion 2021-10-13 (Actual)

PRIMARY OUTCOMES:
safety and tolerability: percentage of patients experiencing treatment-related and treatment-emergent adverse events | up to 5 years
  The percentage of patients experiencing treatment-related and treatment-emergent adverse events
maximum tolerated dose | up to 5 years
  To identify the maximum tolerated dose (MTD) of SL-801 or determine the maximum tested dose at which multiple dose-limiting toxicities (DLTs) are not observed.

SECONDARY OUTCOMES:
Duration of Response | up to 5 years
  to evaluate the duration of response
Progression Free Survival | up to 5 years
  to evaluate progression free survive
Overall Response Rate | up to 5 years
  to evaluate overall response rate
Overall Survival | up to 5 years
  to evaluate overall survival
Pharmacokinetic Profile | up to 5 years
  Determine the maximum concentration of SL-801 in plasma

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Yale Cancer Center, New Haven, Connecticut
  - Florida Cancer Specialist, Sarasota, Florida
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Mary Crowely Cancer Research Centers- Medical City, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Washington, Seattle Cancer Care Alliance, Seattle, Washington

REFERENCES:
- [Background] Ahn C. An evaluation of phase I cancer clinical trial designs. Stat Med. 1998 Jul 30;17(14):1537-49. doi: 10.1002/(sici)1097-0258(19980730)17:143.0.co;2-f. PMID 9699228
- [Background] Arnaoutov A, Azuma Y, Ribbeck K, Joseph J, Boyarchuk Y, Karpova T, McNally J, Dasso M. Crm1 is a mitotic effector of Ran-GTP in somatic cells. Nat Cell Biol. 2005 Jun;7(6):626-32. doi: 10.1038/ncb1263. PMID 15908946
- [Background] Dillman RO, Koziol JA. Phase I cancer trials: limitations and implications. Mol Biother. 1992 Sep;4(3):117-21. PMID 1445664
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Background] Gatsonis C, Greenhouse JB. Bayesian methods for phase I clinical trials. Stat Med. 1992 Jul;11(10):1377-89. doi: 10.1002/sim.4780111011. PMID 1518998
- [Background] Gerecitano J. SINE (selective inhibitor of nuclear export)--translational science in a new class of anti-cancer agents. J Hematol Oncol. 2014 Oct 4;7:67. doi: 10.1186/s13045-014-0067-3. PMID 25281264
- [Background] Huang WY, Yue L, Qiu WS, Wang LW, Zhou XH, Sun YJ. Prognostic value of CRM1 in pancreas cancer. Clin Invest Med. 2009 Dec 1;32(6):E315. PMID 20003838
- [Background] International Conference on Harmonisation. E8: General Considerations for Clinical Trials, July 1997.
- [Background] Kojima K, Kornblau SM, Ruvolo V, Dilip A, Duvvuri S, Davis RE, Zhang M, Wang Z, Coombes KR, Zhang N, Qiu YH, Burks JK, Kantarjian H, Shacham S, Kauffman M, Andreeff M. Prognostic impact and targeting of CRM1 in acute myeloid leukemia. Blood. 2013 May 16;121(20):4166-74. doi: 10.1182/blood-2012-08-447581. Epub 2013 Apr 5. PMID 23564911
- [Background] Lapalombella R, Sun Q, Williams K, Tangeman L, Jha S, Zhong Y, Goettl V, Mahoney E, Berglund C, Gupta S, Farmer A, Mani R, Johnson AJ, Lucas D, Mo X, Daelemans D, Sandanayaka V, Shechter S, McCauley D, Shacham S, Kauffman M, Chook YM, Byrd JC. Selective inhibitors of nuclear export show that CRM1/XPO1 is a target in chronic lymphocytic leukemia. Blood. 2012 Nov 29;120(23):4621-34. doi: 10.1182/blood-2012-05-429506. Epub 2012 Oct 3. PMID 23034282
- [Background] Lassen UN, Mau-Soerensen M, Kung AL, Wen PY, Lee EQ, Plotkin SR, et al. A phase 2 study on efficacy, safety and intratumoral pharmacokinetics of oral selinexor (KPT-330) in patients with recurrent glioblastoma (GBM). J Clin Oncol 33, 2015 (suppl; abstr 2044)
- [Background] Noske A, Weichert W, Niesporek S, Roske A, Buckendahl AC, Koch I, Sehouli J, Dietel M, Denkert C. Expression of the nuclear export protein chromosomal region maintenance/exportin 1/Xpo1 is a prognostic factor in human ovarian cancer. Cancer. 2008 Apr 15;112(8):1733-43. doi: 10.1002/cncr.23354. PMID 18306389
- [Background] Pathria G, Wagner C, Wagner SN. Inhibition of CRM1-mediated nucleocytoplasmic transport: triggering human melanoma cell apoptosis by perturbing multiple cellular pathways. J Invest Dermatol. 2012 Dec;132(12):2780-90. doi: 10.1038/jid.2012.233. Epub 2012 Jul 26. PMID 22832492
- [Background] Saito N, Sakakibara K, Sato T, Friedman JM, Kufe DW, VonHoff DD, Kawabe T. CBS9106-induced CRM1 degradation is mediated by cullin ring ligase activity and the neddylation pathway. Mol Cancer Ther. 2014 Dec;13(12):3013-23. doi: 10.1158/1535-7163.MCT-14-0064. Epub 2014 Sep 24. PMID 25253782
- [Background] Sakakibara K, Saito N, Sato T, Suzuki A, Hasegawa Y, Friedman JM, Kufe DW, Vonhoff DD, Iwami T, Kawabe T. CBS9106 is a novel reversible oral CRM1 inhibitor with CRM1 degrading activity. Blood. 2011 Oct 6;118(14):3922-31. doi: 10.1182/blood-2011-01-333138. Epub 2011 Aug 12. PMID 21841164
- [Background] Senapedis WT, Baloglu E, Landesman Y. Clinical translation of nuclear export inhibitors in cancer. Semin Cancer Biol. 2014 Aug;27:74-86. doi: 10.1016/j.semcancer.2014.04.005. Epub 2014 Apr 19. PMID 24755012
- [Background] Siddiqui N, Borden KL. mRNA export and cancer. Wiley Interdiscip Rev RNA. 2012 Jan-Feb;3(1):13-25. doi: 10.1002/wrna.101. Epub 2011 Jul 27. PMID 21796793
- [Background] Storer BE. Design and analysis of phase I clinical trials. Biometrics. 1989 Sep;45(3):925-37. PMID 2790129
- [Background] Tan DS, Bedard PL, Kuruvilla J, Siu LL, Razak AR. Promising SINEs for embargoing nuclear-cytoplasmic export as an anticancer strategy. Cancer Discov. 2014 May;4(5):527-37. doi: 10.1158/2159-8290.CD-13-1005. Epub 2014 Apr 17. PMID 24743138
- [Background] Tan DSP, Pang M-Y, Yong WP, Soo RA, Chee CE, Thian YL et al. Phase I study of the safety and tolerability of the Exportin 1 (XPO1) inhibitor Selinexor (SXR) in Asian patients (pts) with advanced solid cancers. J Clin Oncol 33, 2015 (suppl; abstr 2542).
- [Background] Turner JG, Dawson J, Sullivan DM. Nuclear export of proteins and drug resistance in cancer. Biochem Pharmacol. 2012 Apr 15;83(8):1021-32. doi: 10.1016/j.bcp.2011.12.016. Epub 2011 Dec 20. PMID 22209898
- [Background] van der Watt PJ, Maske CP, Hendricks DT, Parker MI, Denny L, Govender D, Birrer MJ, Leaner VD. The Karyopherin proteins, Crm1 and Karyopherin beta1, are overexpressed in cervical cancer and are critical for cancer cell survival and proliferation. Int J Cancer. 2009 Apr 15;124(8):1829-40. doi: 10.1002/ijc.24146. PMID 19117056
- [Background] Walker CJ, Oaks JJ, Santhanam R, Neviani P, Harb JG, Ferenchak G, Ellis JJ, Landesman Y, Eisfeld AK, Gabrail NY, Smith CL, Caligiuri MA, Hokland P, Roy DC, Reid A, Milojkovic D, Goldman JM, Apperley J, Garzon R, Marcucci G, Shacham S, Kauffman MG, Perrotti D. Preclinical and clinical efficacy of XPO1/CRM1 inhibition by the karyopherin inhibitor KPT-330 in Ph+ leukemias. Blood. 2013 Oct 24;122(17):3034-44. doi: 10.1182/blood-2013-04-495374. Epub 2013 Aug 22. PMID 23970380
- [Background] Wang W, Budhu A, Forgues M, Wang XW. Temporal and spatial control of nucleophosmin by the Ran-Crm1 complex in centrosome duplication. Nat Cell Biol. 2005 Aug;7(8):823-30. doi: 10.1038/ncb1282. Epub 2005 Jul 24. PMID 16041368